CLINICAL TRIAL: NCT00719563
Title: The Use of American Ginseng (Panax Quinquefolius) to Improve Cancer-Related Fatigue: A Randomized, Double-Blind, Placebo-Controlled Phase III Study
Brief Title: American Ginseng in Treating Patients With Fatigue Caused by Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NCCTG-N07C2; NCI-2009-00872 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000597665 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2008-07-18; First posted 2008-07-21 (Estimated); Results first posted 2014-08-06 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2016-12

CONDITIONS: Chronic Myeloproliferative Disorders; Fatigue; Leukemia; Lymphoma; Lymphoproliferative Disorder; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms; Precancerous Condition; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: fatigue; unspecified adult solid tumor, protocol specific; accelerated phase chronic myelogenous leukemia; acute undifferentiated leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); atypical chronic myeloid leukemia, BCR-ABL1 negative; blastic phase chronic myelogenous leukemia; chronic myelomonocytic leukemia; chronic phase chronic myelogenous leukemia; mast cell leukemia; progressive hairy cell leukemia, initial treatment; prolymphocytic leukemia; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; recurrent adult T-cell leukemia/lymphoma; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; stage 0 chronic lymphocytic leukemia; stage I adult T-cell leukemia/lymphoma; stage I chronic lymphocytic leukemia; stage II adult T-cell leukemia/lymphoma; stage II chronic lymphocytic leukemia; stage III adult T-cell leukemia/lymphoma; stage III chronic lymphocytic leukemia; stage IV adult T-cell leukemia/lymphoma; stage IV chronic lymphocytic leukemia; T-cell large granular lymphocyte leukemia; untreated adult acute lymphoblastic leukemia; recurrent adult Hodgkin lymphoma; stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; cutaneous B-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent mycosis fungoides/Sezary syndrome; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; adult grade III lymphomatoid granulomatosis; adult nasal type extranodal NK/T-cell lymphoma; Waldenström macroglobulinemia; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult lymphoblastic lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; stage I adult Burkitt lymphoma; stage I adult diffuse large cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I mantle cell lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult grade III lymphomatoid granulomatosis; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; intraocular lymphoma; post-transplant lymphoproliferative disorder; chronic eosinophilic leukemia; chronic neutrophilic leukemia; primary myelofibrosis; essential thrombocythemia; polycythemia vera; extramedullary plasmacytoma; isolated plasmacytoma of bone; monoclonal gammopathy of undetermined significance; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; primary systemic amyloidosis; refractory multiple myeloma; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; myelodysplastic/myeloproliferative neoplasm, unclassifiable
MeSH Terms: conditions — Myeloproliferative Disorders; Fatigue; Leukemia; Lymphoma; Lymphoproliferative Disorders; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Precancerous Conditions; Leukemia, Myeloid, Accelerated Phase; Leukemia, Biphenotypic, Acute; Congenital Abnormalities; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Leukemia, Mast-Cell; Leukemia, Prolymphocytic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Leukemia, Large Granular Lymphocytic; Hodgkin Disease; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Lymphoma, Extranodal NK-T-Cell; Waldenstrom Macroglobulinemia; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Intraocular Lymphoma; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Neutrophilic, Chronic; Primary Myelofibrosis; Thrombocythemia, Essential; Polycythemia Vera; Monoclonal Gammopathy of Undetermined Significance; Immunoglobulin Light-chain Amyloidosis | interventions — Asian ginseng

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive oral American ginseng twice daily for 14 days. Treatment repeats every 2 weeks for 4 courses.
  Interventions: Drug: American ginseng
- Arm II (Placebo Comparator): Patients receive oral placebo twice daily for 14 days. Treatment repeats every 2 weeks for 4 courses.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: American ginseng — Given orally
  Arms: Arm I
Other: placebo — Given orally
  Arms: Arm II

SUMMARY:
RATIONALE: American ginseng may reduce fatigue in patients with cancer. It is not yet known whether American ginseng is more effective than a placebo in treating cancer-related fatigue.

PURPOSE: This randomized phase III trial is studying American ginseng to see how well it works in treating patients with fatigue caused by cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the efficacy of American ginseng (Panax quinquefolius) as therapy for cancer-related fatigue as measured by the general subscale of the Multidimensional Fatigue Symptom Inventory-Short Form (MFSI-SF).

Secondary

* To evaluate toxicities and tolerability of American ginseng when used for cancer-related fatigue.
* To examine stress as a mediating variable on the effects of American ginseng on cancer-related fatigue.
* To explore the impact of American ginseng on various dimensions of fatigue as measured by the other subscales of the MFSI-SF, functional interference as measured by the Brief Fatigue Inventory (BFI), stress as measured by the Perceived Stress Scale, and well being as measured by the Profile of Mood States (POMS), as well as the single measure of fatigue.
* To determine clinically significant changes in fatigue scores using the global impression of change.
* To evaluate whether there are differences in the efficacy of American ginseng for fatigue based on minority populations.

Tertiary

* To describe cortisol and cytokine values in fatigued cancer survivors and to evaluate the relationship of cortisol and cytokines to fatigue severity as well as to patterns of alterations previously documented in fatigued breast cancer survivors.
* To evaluate whether Wisconsin Ginseng impacts the expression of cortisol and cytokine in fatigued cancer survivors.
* To evaluate the role of cortisol and cytokine changes as the mechanism by which Wisconsin Ginseng can ameliorate cancer related fatigue.
* To evaluate the relationships between cytokine and cortisol levels with secondary outcomes such as mood and stress.

OUTLINE: This is a multicenter study. Patients are stratified according to baseline fatigue score (4-7 vs 8-10), disease status of current cancer (initial diagnosis vs recurrent disease), current treatment (chemotherapy, radiation, endocrine therapy [i.e., tamoxifen or aromatase inhibitors], or other targeted therapy) ( yes vs no), duration of all prior cancer treatment in patient's lifetime (none vs ≤ 180 days vs > 180 days), and current tumor type (hematologic vs solid tumor malignancy). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral American ginseng twice daily for 14 days. Treatment repeats every 2 weeks for 4 courses until disease progression or unacceptable toxicity.
* Arm II: Patients receive oral placebo twice daily for 14 days. Treatment repeats every 2 weeks for 4 courses.

Patients are instructed to complete the Ginseng Symptom Experience Diary and the Linear Analogue Scale weekly. Patients also complete the Multidimensional Fatigue Symptom Inventory-Short Form (MFSI-SF), the Profile of Mood States (POMS), and the Brief Fatigue Inventory (BFI) questionnaires at baseline and periodically during study therapy.

Patients who are not actively receiving chemotherapy or radiation therapy undergo blood and saliva sample collection at baseline and periodically during study therapy for correlative studies.

ELIGIBILITY:
1. Required characteristics

   * ≥ 18 years of age
   * Men or women with a history of cancer-related fatigue as defined by an average score ≥ 4 over the past 30 days on the numeric analogue scale (1 - 10)
   * The presence of fatigue ≥ 1 month prior to randomization
   * ECOG performance score 0, 1, or 2
   * Histologic or cytologic proven cancer other than brain cancer or CNS lymphoma, undergoing curative intent therapy (including anti-hormonal therapies such as tamoxifen or leuprolide) or those having completed curative intent therapy who were diagnosed within the past 2 years

     * Note: If a patient is receiving treatment for their disease such as chemotherapy, targeted therapies, immunotherapy or radiation therapy then, the patient must have completed ≥ 1 cycle of chemotherapy, targeted therapy, or ≥ 1 week of radiation treatment.
   * Laboratory values obtained prior to randomization:

     * Hgb ≥ 11 (must be obtained ≤ 30 days; patients must not be transfused ≤ 30 days to meet this criterion)
     * Creatinine ≤ 1.2 x UNL (must be obtained ≤ 180 days prior to randomization)
     * AST (SGOT) or ALT (SGPT) ≤ 1.5 x UNL (must be obtained ≤ 180 days prior to randomization)
   * Negative pregnancy test done ≤ 7 days prior to registration, for women of childbearing potential only
   * Ability to complete patient questionnaires alone or with assistance
   * Controlled:

     * Pain (≤ 4 on Linear Analogue Scale)
     * Insomnia (≤ 4 on Linear Analogue Scale)
   * Willingness to provide blood/saliva samples for correlative studies.

     * Note: These samples are only required for those not receiving active treatment for their disease. Active treatment is defined as chemotherapy, radiation therapy, or immunotherapy, not anti-hormone therapy such as tamoxifen, aromatase inhibitors or leuprolide.
2. Contraindications

   * Hypersensitivity to ginseng
   * Prior use of ginseng capsules for fatigue in the past year

     * Note: Prior use of teas or drinks containing ginseng is allowed, however, patients will be asked to avoid these beverages while on the study.
   * Uncontrolled hypertension on more than one occasion (diastolic blood pressure > 100, systolic > 160) measured ≤ 90 days prior to randomization
   * Currently using any other pharmacologic agents or nonpharmacologic interventions to specifically treat fatigue including psychostimulants, antidepressants, acupuncture, etc.

     * Note: Antidepressants used to treat items other than fatigue (such as hot flashes) are allowed if the patient has been on a stable dose for ≥ 1 month and plans to continue for ≥ 1 month. Erythropoietin agents to treat anemia are allowed. Exercise is allowed.
   * Known brain metastasis or primary CNS malignancy
   * Chronic systemic steroid use (including CHOP therapy or as part of any regular cancer treatment, however, steroids used as prophylaxis for nausea and vomiting are allowed) to prevent rash with Alimta, low dose dexamethasone will be allowed.
   * Diabetes Type I or II (defined by being on oral hypoglycemics or insulin).
   * Psychiatric disorder such as severe depression, manic depressive disorder, obsessive compulsive disorder or schizophrenia. (Defined per medical history).
   * ≤ 4 weeks from major surgery to randomization, including any procedure that requires general anesthetic
   * Any of the following:

     * Pregnant women
     * Nursing women
     * Women of childbearing potential who are unwilling to employ adequate contraception
   * Pain requiring opioid pain medication, however, over the counter analgesics such as Tylenol or ibuprofen are allowed.
   * Use of full dose of anticoagulant therapy (Exception: 1 mg/day of Coumadin for preventing catheter clots is allowed).
   * Use of MAO inhibitors.
   * Planning to start or complete any type of cancer therapy during the 8 week, double blind, course of the study, once randomized on the study. Note: If not currently getting treatment, no chemotherapy agents ≤ 21 days prior to randomization. Combination treatment regimens that have components ending at different times are allowed, as long as any part of the initially started treatment continues through the double blind portion of the study.
   * Malnutrition, active infection, significant pulmonary disease and cardiovascular disease as determined by the physician, as they could impact fatigue.
   * Use of any over the counter herbal/dietary supplement marketed for fatigue or energy (for example, products containing any type of ginseng, rhodiola rosea, high doses of caffeine, guarana, or anything called an "adaptogen").
   * Uncontrolled nausea or vomiting or any symptom that would prevent the ability to comply with daily oral ginseng/placebo treatment.
   * Uncontrolled thyroid disorder.
   * Currently receiving single agent on blinded placebo controlled treatment trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Actual)
Dates: Start 2008-10; Primary Completion 2011-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debra Barton, RN, PhD, AOCN, FAAN, Study Chair — University of Michigan
Locations (326):
- United States (326):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Lusitana, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - Hawaii Medical Center - East, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Kauai Medical Clinic, Lihue, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Pacific Cancer Institute - Maui, Wailuku, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare - Galesburg, Galesburg, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Moline, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - OSF Holy Family Medical Center, Monmouth, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Illinois CancerCare - Spring Valley, Spring Valley, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Michiana Hematology-Oncology, PC - Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - Michiana Hematology Oncology PC - Plymouth, Plymouth, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Michiana Hematology Oncology PC - La Porte, Westville, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Bettendorf, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Hospital District Sixth of Harper County, Anthony, Kansas
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Ochsner Health Center - Bluebonnet, Baton Rouge, Louisiana
  - Ochsner Health Center - Covington, Covington, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - Michiana Hematology Oncology PC - Niles, Niles, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Alexandria, Minnesota
  - MeritCare Bemidji, Bemidji, Minnesota
  - St. Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fergus Falls Medical Group, PA, Fergus Falls, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Immanuel St. Joseph's, Mankato, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Goldschmidt Cancer Center, Jefferson City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Comprehensive Cancer Care, PC, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Lovelace Medical Center - Downtown, Albuquerque, New Mexico
  - Hematology Oncology Associates, PC, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - North Coast Cancer Care - Clyde, Clyde, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Community Cancer Center, Elyria, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - United States Air Force Medical Center - Wright-Patterson, Wright-Patterson AFB, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Willamette Falls Hospital, Oregon City, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - St. Joseph Cancer Center, Bellingham, Washington
  - Cascade Cancer Center at Evergreen Hospital Medical Center, Kirkland, Washington
  - Valley Medical Center, Renton, Washington
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Pacific Medical Center, Seattle, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Edwards Comprehensive Cancer Center at Cabell Huntington Hospital, Huntington, West Virginia
  - Marshfield Clinic - Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Luther Midlelfort Hospital, Eau Claire, Wisconsin
  - Midelfort Clinic - Luther, Eau Claire, Wisconsin
  - Central Wisconsin Cancer Program at Agnesian HealthCare, Fond du Lac, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Franciscan Skemp Healthcare - La Crosse Campus, La Crosse, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - St. Nicholas Hospital, Sheboygan, Wisconsin
  - Marshfield Clinic at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Door County Cancer Center at Door County Memorial Hospital, Sturgeon Bay, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Result] Barton DL, Liu H, Dakhil SR, et al.: Phase III evaluation of American ginseng (panax quinquefolius) to improve cancer-related fatigue: NCCTG trial N07C2. [Abstract] J Clin Oncol 30 (Suppl 15): A-9001, 2012.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three-hundred and sixty-four participants were recruited between October 2008 and July 2011 from 40 North Central Cancer Treatment Group (NCCTG) member sites.
Pre-assignment Details: There were a total of 23 cancellations (12 Ginseng, 11 Placebo) and these 23 patients were excluded from all analysis.
Groups:
- Ginseng: Patients received oral American ginseng twice daily for 14 days. This treatment was repeated every two weeks for 4 courses, for a total of 8 weeks of treatment.
- Placebo: Patients received oral placebo twice daily for 14 days. This treatment was repeated every two weeks for 4 courses, for a total of 8 weeks of treatment.
Period: Overall Study
Arm/Group | Ginseng | Placebo
Started | 171 | 170
Completed | 133 | 128
Not Completed | 38 | 42
Not completed — Adverse Event | 16 | 13
Not completed — Medical condition changed | 3 | 5
Not completed — Lack of Efficacy | 3 | 7
Not completed — Personal reasons | 6 | 7
Not completed — Unknown reasons | 4 | 6
Not completed — Noncompliant | 1 | 1
Not completed — Lost to Follow-up | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ginseng | Placebo | Total
Number analyzed (Participants) | 171 | 170 | 341
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (12.7) | 55.9 (11.8) | 55.6 (12.2)
Gender [Count of Participants; unit: Participants]
  Female | 138 | 128 | 266
  Male | 33 | 42 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 164 | 166 | 330
  Unknown or Not Reported | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 10 | 8 | 18
  White | 155 | 157 | 312
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 171 | 170 | 341
Menopausal status [Number; unit: participants]
  Pre | 37 | 31 | 68
  Post/natural-surgical | 95 | 90 | 185
  Not applicable (Male) | 33 | 42 | 75
  Unknown | 6 | 7 | 13
Time since current cancer diagnosis [Number; unit: participants]
  <180 days | 63 | 64 | 127
  180-360 days | 47 | 42 | 89
  >360 days | 61 | 64 | 125
More than one primary cancer [Number; unit: participants]
  Yes | 40 | 36 | 76
  No | 131 | 134 | 265
Type of cancer [Number; unit: participants]
  Breast | 110 | 96 | 206
  Colon | 20 | 17 | 37
  Prostate | 6 | 8 | 14
  Hematologic | 8 | 9 | 17
  Gynecologic | 5 | 7 | 12
  Combination/unknown/other | 22 | 33 | 55
Currently receiving treatment [Number; unit: participants]
  Yes | 83 | 83 | 166
  No | 88 | 87 | 175
Current endocrine therapy [Number; unit: participants]
  Tamoxifen | 23 | 22 | 45
  Aromatase inhibitor | 27 | 33 | 60
  Antiandrogen | 2 | 5 | 7
  Other | 7 | 3 | 10
  None | 112 | 107 | 219
Sleep aids [Number; unit: participants]
  Yes | 43 | 29 | 72
  No | 128 | 141 | 269
If taking sleep aids, how frequent? [Number; unit: participants]
  Daily | 18 | 16 | 34
  Intermittent | 25 | 13 | 38
  Not taking sleep aids | 128 | 141 | 269
Exercising regularly [Number; unit: participants]
  Yes | 71 | 68 | 139
  No | 98 | 98 | 196
  Missing | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 4 in the General Subscale of the MFSI-SF
Description: Multidimensional Fatigue Symptom Inventory-Short Form (MFSI-SF) general subscale is a six-item subscale to measure the subjective experience of fatigue. The items include feeling "pooped, worn out, fatigued, sluggish, run down and tired". Answers are on a 5-point scale, ranging from 0 (not at all) to 4 (extremely). The subscale scores were the sum of all six items. The scores were converted to a 100-point scale, with higher numbers indicating less fatigue. Change from baseline to week 4 was calculated by subtracting the baseline scores from the scores at week 4.
Time Frame: Baseline and week 4
Population: Includes all participants who completed both baseline and week 4 assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ginseng | Placebo
Number analyzed (Participants) | 147 | 153
units on a scale | 14.4 (27.1) | 8.2 (24.8)
Statistical Analysis 1: Comparison: Ginseng vs Placebo; Test type: Superiority or Other; p = 0.0737, Wilcoxon Rank Sum

2. Secondary Outcome: Number of Treatment Related Grade 2 to 3 Adverse Events >=1% Incidence
Description: Adverse events were assessed by Common Terminology Criteria for Adverse Events (CTCAE) v3.0. Grading: Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe, Grade 4=Life-threatening, Grade 5=Death.
Time Frame: Week 1 to Week 8
Population: Includes all participants that reported at least one value after baseline.
Measure: Number; unit: participants
Arm/Group | Ginseng | Placebo
Number analyzed (Participants) | 168 | 169
participants
  Grade 2 Nausea | 5 | 3
  Grade 2 Vomiting | 2 | 2
  Grade 2 Insomnia | 9 | 10
  Grade 3 Insomnia | 1 | 1
  Grade 2 Anxiety | 4 | 5
  Grade 2 Agitation | 2 | 4

3. Secondary Outcome: Change From Baseline to Week 4 in the Impact on Physical, Mental, and Emotional States and Vigor as Measured by Other Subscales of the MFSI-SF
Description: Each MFSI-SF subscale consist of 6 items on a 5-point scale, ranging from 0 (not at all) to 4 (extremely). The subscale scores were the sum of all six items. The scores were then converted to a 100-point scale, with higher numbers indicating less fatigue. Change from baseline to week 4 was calculated by subtracting the baseline scores from the scores at week 4.
Time Frame: Baseline and Week 4
Population: Includes all participants who completed both baseline and week 4 assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ginseng | Placebo
Number analyzed (Participants) | 147 | 152
units on a scale
  Physical | 1.6 (15.9) | -0.4 (14.7)
  Mental | 2.0 (15.2) | 0.6 (16.1)
  Emotional | 0.5 (16.1) | 0.5 (16.7)
  Vigor | 1.8 (19.0) | 0.4 (15.5)

4. Secondary Outcome: Change From Baseline to Week 4 Fatigue as Measured by the BFI and Linear Analogue Scale of Fatigue
Description: Brief Fatigue Inventory (BFI) consist of 3 items that assess the severity of fatigue and 6 items that assess the impact of fatigue on daily functioning in a 10-points scale with 0 as no fatigue or does not interfere with daily functioning and 10 as bad fatigue or completely interferes. The scores for the six items were summed up to form a total interference score. The linear analogue scale of fatigue was a 10-points scale with 0 as no fatigue and 10 as bad fatigue. All scores were then transformed into 0 to 100 scale, with 100 as less fatigue/less interference. Change from baseline to week 4 was calculated by subtracting the baseline scores from the scores at week 4.
Time Frame: Baseline and Week 4
Population: Includes all participants who completed both baseline and week 4 assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ginseng | Placebo
Number analyzed (Participants) | 150 | 150
units on a scale
  Fatigue Usual | 11.9 (25.7) | 9.9 (23.4)
  Fatigue Now | 11.8 (26.4) | 7.9 (24.1)
  Fatigue Worst | 11.8 (25.6) | 9.7 (25.3)
  BFT Total Interference | 9.2 (22.0) | 5.8 (21.1)

5. Secondary Outcome: Change From Baseline to Week 4 Vigor/Activity and Fatigue-inertia as Measured by POMS
Description: Profile of Mood States (POMS) measures a variety of mood states including tension/anxiety, depression/dejection, anger/hostility, vigor/activity, fatigue/inertia and confusion/bewilderment. Each subscale consist of 5 items with a 5 points-scale (0=not at all, 1=a little, 2=moderately, 3=quite a bit and 4=extremely). The subscale scores were the sum of all five items. The scores were then transformed into a 100-point scale with higher numbers indicating less fatigue. Change from baseline to week 4 was calculated by subtracting the baseline scores from the scores at week 4.
Time Frame: Baseline and Week 4
Population: Includes all participants who completed both baseline and week 4 assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ginseng | Placebo
Number analyzed (Participants) | 139 | 142
units on a scale
  Vigor/Activity | 5.0 (18.7) | 3.9 (17.3)
  Fatigue/Inertial | 14.5 (25.0) | 7.7 (23.6)

6. Secondary Outcome: Change From Baseline to Week 4 for the Impact on Stress as Measured by Perceived Stress Scale (PSS)
Description: PSS consist of 14 items that assess the impact on stress in a 5-points scale (0=never, 1=almost never, 2=sometimes, 3=fairly often and 4=very often). The total scores were the sum of all 14 items. The scores were then transformed into a 100-point scale with higher numbers indication less stress. Change from baseline to week 4 was calculated by subtracting the baseline scores from the scores at week 4.
Time Frame: Baseline and Week 4
Population: Includes all participants who completed both baseline and week 4 assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ginseng | Placebo
Number analyzed (Participants) | 148 | 148
units on a scale | -3.1 (11.1) | -3.2 (10.5)

7. Secondary Outcome: Change From Baseline to Week 8 in the Impact on General, Physical, Mental, and Emotional States and Vigor as Measured by Other Subscales of the MFSI-SF
Description: Each MFSI-SF subscale consist of 6 items on a 5-point scale, ranging from 0 (not at all) to 4 (extremely). The subscale scores were the sum of all six items. The scores were then converted to a 100-point scale, with higher numbers indicating less fatigue. Change from baseline to week 8 was calculated by subtracting the baseline scores from the scores at week 8.
Time Frame: Baseline and week 8
Population: Includes all participants who completed both baseline and week 8 assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ginseng | Placebo
Number analyzed (Participants) | 138 | 133
units on a scale
  General | 20 (27.0) | 10.3 (26.1)
  Physical | 3.0 (17.9) | -1.7 (18.2)
  Mental | 2.8 (16.5) | 3.4 (15.2)
  Emotional | 3.0 (17.4) | 2.3 (17.4)
  Vigor | 4.6 (20.5) | 2.5 (17.6)

8. Secondary Outcome: Change From Baseline to Week 8 Fatigue as Measured by the BFI and Linear Analogue Scale of Fatigue
Description: Brief Fatigue Inventory (BFI) consist of 3 items that assess the severity of fatigue and 6 items that assess the impact of fatigue on daily functioning in a 10-points scale with 0 as no fatigue or does not interfere with daily functioning and 10 as bad fatigue or completely interferes. The scores for the six items were summed up to form a total interference score. The linear analogue scale of fatigue was a 10-points scale with 0 as no fatigue and 10 as bad fatigue. All scores were then transformed into 0 to 100 scale, with 100 as less fatigue/less interference. Change from baseline to week 8 was calculated by subtracting the baseline scores from the scores at week 8.
Time Frame: Baseline and Week 8
Population: Includes all participants who completed both baseline and week 8 assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ginseng | Placebo
Number analyzed (Participants) | 138 | 136
units on a scale
  Fatigue Usual | 16.4 (23.9) | 11.5 (23.8)
  Fatigue Now | 17.6 (27.1) | 8.1 (26.7)
  Fatigue Worst | 16.6 (27.2) | 10.0 (26.9)
  BFI Total Interference | 12.9 (25.6) | 9.0 (23.0)

9. Secondary Outcome: Change From Baseline to Week 8 Vigor/Activity and Fatigue-inertia as Measured by POMS
Description: Profile of Mood States (POMS) measures a variety of mood states including tension/anxiety, depression/dejection, anger/hostility, vigor/activity, fatigue/inertia and confusion/bewilderment. Each subscale consist of 5 items with a 5 points-scale (0=not at all, 1=a little, 2=moderately, 3=quite a bit and 4=extremely). The subscale scores were the sum of all five items. The scores were then transformed into a 100-point scale with higher numbers indicating less fatigue. Change from baseline to week 8 was calculated by subtracting the baseline scores from the scores at week 8.
Time Frame: Baseline and week 8
Population: Includes all participants who completed both baseline and week 8 assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ginseng | Placebo
Number analyzed (Participants) | 132 | 128
units on a scale
  Vigor/Activity | 8.2 (19.8) | 6.4 (19.8)
  Fatigue/Inertia | 18.6 (24.8) | 10.2 (26.1)

10. Secondary Outcome: Change From Baseline to Week 8 for the Impact on Stress as Measured by Perceived Stress Scale (PSS)
Description: PSS consist of 14 items that assess the impact on stress in a 5-points scale (0=never, 1=almost never, 2=sometimes, 3=fairly often and 4=very often). The total scores were the sum of all 14 items. The scores were then transformed into a 100-point scale with higher numbers indication less stress. Change from baseline to week 8 was calculated by subtracting the baseline scores from the scores at week 8.
Time Frame: Baseline and Week 8
Population: Includes all participants who completed both baseline and week 8 assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ginseng | Placebo
Number analyzed (Participants) | 138 | 131
units on a scale | -5.2 (11.7) | -4.7 (10.8)

11. Secondary Outcome: Average Change From Baseline to Week 4 in Fatigue for Those Who Perceive a Change of +2 and +3
Description: Changes in fatigue as measured using subscales of MFSI-SF, the interference scale of the BFI and the linear analogue scale (LASA) fatigue question were compared between arms for those participants who express a perceived change in fatigue via the global impression score of a +2 (moderately better) and +3 (very much better).
Time Frame: Baseline and Week 4
Population: Includes all participants who completed both baseline and week 4 assessments with a perceived change in fatigue via the global impression score of a +2 and +3 at week 4.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ginseng | Placebo
Number analyzed (Participants) | 25 | 24
units on a scale
  MFSI-SF General | 38.8 (23.3) | 29.2 (21.5)
  MFSI-SF Physical | 12.2 (18.3) | 5.7 (15.1)
  MFSI-SF Mental | 8.9 (18.8) | 2.6 (14.9)
  MFSI-SF Emotional | 8.0 (14.4) | 8.7 (16.8)
  MFSI-SF Vigor | 13.4 (22.6) | 12.0 (13.8)
  BFI Total Interference | 27.3 (23.7) | 22.3 (15.2)
  LASA Fatigue | 40.9 (27.0) | 37.0 (19.0)

12. Secondary Outcome: Average Change From Baseline to Week 8 in Fatigue for Those Who Perceive a Change of +2 and +3
Description: Changes in fatigue as measured using subscales of MFSI-SF, the interference scale of the BFI and the linear analogue scale fatigue question were compared between arms for those participants who express a perceived change in fatigue via the global impression score of a +2 (moderately better) and +3 (very much better).
Time Frame: Baseline and Week 8
Population: Includes all participants who completed both baseline and week 8 assessments with a perceived change in fatigue via the global impression score of a +2 and +3 at week 8.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ginseng | Placebo
Number analyzed (Participants) | 34 | 35
units on a scale
  MFSI-SF General | 35.7 (24.7) | 30.6 (22.5)
  MFSI-SF Physical | 7.6 (17.5) | 3.8 (20.8)
  MFSI-SF Mental | 5.3 (19.0) | 5.3 (16.1)
  MFSI-SF Emotional | 9.8 (14.8) | 9.8 (15.9)
  MFSI-SF Vigor | 18.0 (18.5) | 12.6 (13.2)
  BFI Total Interference | 30.6 (23.5) | 20.9 (20.5)
  LASA Fatigue | 41.8 (19.5) | 38.1 (18.3)

13. Secondary Outcome: Change From Baseline to Week 4 in the General Subscale of the MFSI-SF for Minority Populations
Description: as for outcome 1
Time Frame: Baseline and Week 4
Population: The analysis was not able to be done due to the low numbers of minorities accrued.
Arm/Group | Ginseng | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Ginseng | Placebo
Serious Adverse Events (participants affected / at risk) | 1/168 | 5/169
Other Adverse Events (participants affected / at risk) | 115/168 | 112/169
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ginseng (N=168) | Placebo (N=169)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ginseng (N=168) | Placebo (N=169)
Hemoglobin decreased (Blood and lymphatic system disorders) | 2 (3) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (4) | 0 (0)
Dry eye syndrome (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colonic obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (2)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (2)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 55 (119) | 51 (101)
Tooth disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 12 (18) | 22 (33)
Fatigue (General disorders) | 3 (4) | 4 (6)
Fever (General disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Leukocyte count decreased (Investigations) | 4 (6) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 6 (9) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 28 (54) | 37 (96)
Anxiety (Psychiatric disorders) | 40 (84) | 45 (110)
Insomnia (Psychiatric disorders) | 80 (205) | 82 (218)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 3 (7)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes